CLINICAL TRIAL: NCT03062332
Title: Altered Fecal Microbiota Composition in Patients With Major Depressive Disorder and Bipolar Disorder
Brief Title: The Gut Microbiota of Bipolar and Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: TGMOBAD2017
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Bipolar disorder,mania: The group includes subjects who are diagnosed to mania episode of bipolar disorder.
  Interventions: Genetic: Faecal genome
- Bipolar disorder,depressive: The group includes subjects who are diagnosed to depression episode of bipolar disorder.
  Interventions: Genetic: Faecal genome
- Bipolar disorder,mixed: The group includes subjects who are diagnosed to mixed episode of bipolar disorder.
  Interventions: Genetic: Faecal genome
- First episode major depression: The group includes subjects who are diagnosed to first episode of major depression.
  Interventions: Genetic: Faecal genome
- major depression，recurrent: The group includes subjects who are diagnosed to recurrent episode of major depression.
  Interventions: Genetic: Faecal genome
- Healthy control: The group includes subjects who are Healthy control.
  Interventions: Genetic: Faecal genome

INTERVENTIONS:
Genetic: Faecal genome — Sequencing faecal genome is not the intervention measure.It is the Observational method to detect the component of faecal microbiota.

SUMMARY:
Background: The gut microbiome is emerging as an important factor in regulating mental health yet it remains unclear what the target should be for psychiatric treatment. Investigators aim at elucidating the complement of the gut microbiome community for individuals with Major Depressive disorder (MDD) and Bipolar disorder (BD) relative to controls, and test for relationships with symptoms.

Methods: Investigators prospect to recruit subjects including patients and controls amount to 240. All subjects will be collected for blood and stool samples,assessed by clinical scales. Finally, analyzing the correlation among the metabolon in blood, microbiota in stool and clinical scales to obtain the possible interaction between diseases and gut microbiota.

DETAILED DESCRIPTION:
Background: MDD (Major Depressive disorder) and BD (Bipolar disorder), whose specific pathogenesis is still unclear, are both a multi-factorial disease being caused by biological, psychological and social factors. Accumulating evidence suggests that gut microbiota play an important role in brain functions and in the pathogenesis of neuropsychiatric diseases, such as autism, anxiety, as well as depression. No study has thus far compared the human gut microbiota among BD, MDD and the healthy control (HC). The aim of this study is to compare the composition of fecal microbiota among BD, MDD and HC. Furthermore, investigators aim at identifying direct correlations between human fecal microbiota (as a proxy for gut microbiota) and symptoms.

Methods:

1. Investigators aim at recruiting human subjects in total 240, which including mania episode of bipolar disorder (40), depressive episode of bipolar disorder (40), mixed episode of bipolar disorder (40), first episode of major depressive disorder (40), recurrent episode of major depressive disorder (40), and healthy control (40). All patients, diagnosed according to the research criteria of the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10）, come from The First Affiliated Hospital of Xi'an Jiaotong University and controls are healthy volunteers.
2. Collecting blood and stool samples, evaluating clinical scales including Montgomery-Asberg Depression Scale (MADRS), Young Mania Rating Scale (YMRS), Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAMA), Measurement And Treatment Research To Improve Cognition In Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB), Clinical Global Impression (CGI) are all finished in first day after threshold.
3. Measure the metabolon in blood such as S-CFA, and gut microbiota.
4. Using Statistical Program for Social Sciences (SPSS) to compare general and clinical data among groups and analyze the correlation between the microbiota and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Conforms to the diagnosis of bipolar disorder or major depressive disorder.
* Take antibiotics continuously less than 3 days in recent 3 months.
* 17.5≦BMI≦30
* Age≦65

Exclusion Criteria:

* who is diagnosed with physical diseases and other mental diseases.
* pregnant or lactational women
* who is diagnosed with mental retardation.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are someone who are hospitalized in First Affiliated Hospital of Xi'an Jiaotong University.
  Healthy controls are healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Composition of the gut microbiota | 3 months
  The relative richness of the species, %

SECONDARY OUTCOMES:
metabolon | 3 months
  the concentration of short-chain fatty acid(S-CFA), μg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Xiancang Ma, professor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Xiancang Ma, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No